CLINICAL TRIAL: NCT00176787
Title: Phase II Trial of Preoperative Radiation Therapy With Capecitabine in Rectal Cancer (UMCC 0046)
Brief Title: Radiation Therapy With Capecitabine in Rectal Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: recruitment goals met
Sponsor: University of Michigan Rogel Cancer Center (Other)
Collaborators: Hoffmann-La Roche (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UMCC 0046
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Last update posted 2008-01-10 (Estimated); Status verified 2007-12

CONDITIONS: Rectal Cancer
MeSH Terms: conditions — Rectal Neoplasms | interventions — Capecitabine; Radiation; Surgical Procedures, Operative

INTERVENTIONS:
Drug: Capecitabine
Procedure: Radiation
Procedure: Surgery

SUMMARY:
This study will use an experimental combination of treatment with the drug Capecitabine and radiation therapy prior to an operation for removal of the patient's tumor. The drug Capecitabine is an oral form of a drug called 5-FU which has been widely used to treat rectal cancer.

This is a phase II clinical trial, which means that the physician will be studying the reactions of the patient's body and tumor to treatment with Capecitabine and radiation therapy. The purpose of this study is to see if the tumor responds to this treatment and to determine how long the response lasts. The study also will see what kind of side effects this experimental treatment causes and see how often these side effects occur.

Preliminary human studies using Capecitabine and radiation therapy have produced encouraging results with acceptable side effects.

ELIGIBILITY:
Eligibility Criteria

1. Histologic confirmation of adenocarcinoma of the rectum.
2. The lesion must be located in the rectum. For purposes of this study, the lesion must be within 12 cm of the anus as measured by sigmoidoscopy.
3. Patients must have indication of a locally advanced lesion defined for this study as tumor through the bowel wall (> T3) or involving regional lymph nodes (>N1). Clinical stage determination may be made by physical examination (for T4 lesions only), endoscopic ultrasound or CT scan of pelvis.
4. Patients with metastatic disease are eligible provided operative intervention on primary site is anticipated.
5. Patients must have adequate organ function defined as pretreatment leukocyte count > 3,000/ul, platelet count > 100,000/ul, serum creatinine < 2.0 mg/dl, serum bilirubin < 2 mg/dl. Note: Capecitabine is contraindicated in patients with severe renal impairment (creatinine clearance < 30 ml/min). In patients with calculated creatinine clearance of 30-50 ml/min capecitabine will begin at (-)1 level dose reduction (see section 6.3)
6. Patients must be at least 18 years of age and have a Zubrod performance status of < 2 (see appendix 1.)
7. Patients must be informed of the investigational nature of this study and provide written informed consent in accordance with institutional and federal guidelines prior to the initiation of therapy.

Exclusion Criteria:

1. Patients may not have received previous pelvic irradiation for any indication, or previous chemotherapy for cancer therapy within the preceding 6 months.
2. Patients must have no other serious medical or psychiatric illness that would limit the ability of the patient to receive protocol therapy or provide informed consent.
3. Pregnant or lactating women may not participate. Women/men of reproductive potential must agree to use an effective contraceptive method.
4. Patients with lack of physical integrity of the upper gastrointestinal tract, inability to swallow tablets or those who have malabsorption syndrome are not eligible.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30
Dates: Start 2000-10; Primary Completion 2005-05 (Actual); Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
Objectives:
In patients with locally advanced rectal cancer treated with preoperative radiation and capecitabine chemotherapy to estimate:
a. the pathologic complete response rate
b. the clinical response rate
c. the proportion of patients converted to sphincter sparing surgery
clinical response rate | 2 cycles
d. The quantitative and qualitative toxicities of the treatment approach
e. The relationship of intratumoral levels of thymidylate synthase, dipyrimidine dehydrogenase and thymidine phosphorylase determined immunohistochemically to response

CONTACTS AND LOCATIONS:
Overall Officials: Mark Zalupski, M.D., Principal Investigator — University of Michigan Rogel Cancer Center
Locations (1):
- University of Michigan Cancer Center, Ann Arbor, Michigan, United States